CLINICAL TRIAL: NCT05809570
Title: Periodontal Disease Prediction System and a Patient-Specific Gingival Recession Simulator
Brief Title: Periodontal Disease Prediction System
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Abant Izzet Baysal University (Other); Istanbul Technical University (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Şadiye GÜNPINAR, Principal Investigator, Bezmialem Vakif University
Other Study IDs: 119S025
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Periodontal Diseases
Keywords: gingival recession; Oral hygiene motivation; Computer-aided design
MeSH Terms: conditions — Periodontal Diseases; Gingival Recession | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Periodontal examination: Cross- sectional clinical periodontal examinations and measurements were performed using a Williams periodontal probe
  Interventions: Diagnostic Test: Clinical examination

INTERVENTIONS:
Diagnostic Test: Clinical examination — A total of 1057 individuals who applied to Bolu Abant İzzet Baysal University, Faculty of Dentistry, Department of Periodontology and agreed to participate in the study were clinically and radiologically examined.
  An intraoral scanner was utilized to capture direct optical intraoral data of a patient.

SUMMARY:
The purpose of this study was to develop a periodontal disease prediction software and a patient-based gingival recession simulator for clinical practice aiming at improving oral hygiene motivation of patients with periodontal problems.

DETAILED DESCRIPTION:
Periodontal Disease Prediction (PDP) software has three components: a) Data Loading Window (DLW) b) Three-Dimensional Mouth Model (3DM) and c) Periodontal Attachment Loss Indicator (PLI). Demographic and clinical examinations of 1057 volunteers were recorded to DLW. An unsupervised machine learning K means clustering analysis was used to categorize the data obtained from the study population and identified the periodontal risk groups. An intraoral scanner was utilized to capture direct optical intraoral data of a patient and transferred to the 3DM. The intraoral model went under two algorithm steps for obtaining a recessed model. First, gingival curves separating gingiva and tooth were extracted using a Dijkstra's algorithm. Limit curves determining boundaries of recessed regions in the intraoral model were then obtained using gingival curves. The gingival recession was then mimicked by losing gingiva and disappearing tooth roots at proper locations in the intraoral model and Additionally, the final four different 3 dimensional recessed model (maxilla, mandibula, anterior teeth and posterior teeth) belonging to the same patient were scored based on the similarity to the real gingival recession by 25 periodontology specialist via online survey.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years,
* Periodontal status ranging from no clinical periodontal disease (<10% with bleeding on probing) to periodontitis (stage I to IV)
* Patients having at least one teeth in each quadrant were included.

Exclusion Criteria:

* Patients undergoing orthodontic treatment and using anti-inflammatory drugs were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who applied to Bolu Abant İzzet Baysal University, Faculty of Dentistry, Department of Periodontology for their rutin periodontal controls or complains about gingival problems were included in this study.
Sampling Method: Probability Sample
Enrollment: 1057 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Number of sites Clinical Attachment Loss≥5 mm | Baseline
  Categorized as: None, <4, 4-8, >8

SECONDARY OUTCOMES:
Presence of diabetes | Baseline
  Categorized as: Absence, diabetes with HbA1c<7, diabetes with HbA1c≥7
Smoking status | Baseline
  Categorized as: None, < 10 per day, ≥10 per day
Patient cooperation and awareness | Baseline
  Categorized as: None, some, high
History of dental treatment | Baseline
  Categorized as: None, treated in the last 1 year
Tooth brushing Habits | Baseline
  Categorized as: None/ 1 time in day/ ≥2 times in day
Interproximal cleaning | Baseline
  Categorized as: None/ 1 time in day/ ≥2 times in day
Alveolar bone loss/age | Baseline
  Categorized as: None/ <0.25 /0.25-1/ >1
Number of sites Probing Pocket Depth ≥5 mm | Baseline
  Categorized as: None/ <4 / 4-8/ >8
Number of sites Bleeding on Probing (%) | Baseline
  Categorized as: <10%/ 10-25%/ >25%
Tooth mobility | Baseline
  Categorized as: None/ Miller I/ Miller II/ Miller III
Gingival phenotype | Baseline
  Categorized as: Thin/thick
Presence of furcation involvement | Baseline
  Categorized as: None/ horizontal involvement/ vertical involvement/ combined
Vertical alveolar bone loss | Baseline
  Categorized as: Presence/absence
Presence of endodontic tooth problem | Baseline
  Categorized as: Presence/absence
Number of tooth loss | Baseline
  Categorized as: None/ <4/ 4-8/ >8
Traumatic occlusion | Baseline
  Categorized as: Presence/absence
Restorations including gingival margin | Baseline
  Categorized as: Presence/absence

CONTACTS AND LOCATIONS:
Overall Officials: Şadiye Günpınar, Assoc. Prof, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared if the researchers contact to the principal investigator after 6 months following the publication